CLINICAL TRIAL: NCT01079715
Title: Safety and Efficacy of Treatment With Propranolol in Newborns With Retinopathy of Prematurity: a Pilot Study
Brief Title: Safety and Efficacy of Propranolol in Newborns With Retinopathy of Prematurity
Acronym: PROP-ROP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Collaborators: Ospedale Maggiore Policlinico Mangiagalli e Regina Elena (Other)
Responsible Party: Principal Investigator, Luca Filippi, Dr. Luca Filippi, Meyer Children's Hospital IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EudraCT Number 2010-018737-21
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Retinopathy of Prematurity
Keywords: Newborn; Retinal Diseases; Angiogenesis Modulating Agents; Adrenergic beta-Antagonists
MeSH Terms: conditions — Retinopathy of Prematurity; Retinal Diseases | interventions — Propranolol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propranolol (Experimental): Oral Propranolol administration is the experimental arm of this study
  Interventions: Drug: Propranolol
- Control (No Intervention): Control arm is treated following the standard treatment schedule of Early Treatment For Retinopathy Of Prematurity Cooperative Group

INTERVENTIONS:
Drug: Propranolol — Dosage of 0.5mg/Kg oral, every 6 hours. The study will be discontinued immediately in the presence of serious adverse effects attributable to the pharmacological actions of propranolol (severe hypotension, bradycardia or bronchospasm).
  In case such events occur in any of the 3 groups of gestational age, the study could start again with half dose (0.25mg/Kg oral, every 6 hours) after notification to the Ethics Committee.
  In case of surgery or induction of anesthesia during the administration of propranolol, the drug should be discontinued at least 24 hours before surgery.
  In cases of severe hypotension or bradycardia may be administered one or more of the following drugs:
  * Atropine.
  * Isoproterenol hydrochloride (isoprenaline.
  * Terlipressin.
  * Glucagon In case of severe bronchospasm may be used salbutamol aerosol or salbutamol + ipratropium bromide. Betamethasone could be used for aerosol or systemic (intravenous or intramuscular).
  Arms: Propranolol

SUMMARY:
The purpose of this study is to determine whether the administration of propranolol is effective in the treatment of the retinopathy of the prematurity.

DETAILED DESCRIPTION:
Retinopathy of Prematurity (ROP) is still a major cause of blindness in children in developed countries around the world, and an increasing cause of blindness in developing countries. The ablation of the retina with photocoagulation by laser or cryotherapy reduces the incidence of blindness by suppressing the neovascular phase of ROP. However, the visual outcomes after treatment are often poor. The development of ROP depends largely from vascular endothelial growth factor (VEGF). The reduction of VEGF expression in the neovascular phase might prevent destructive neovascularization in ROP.

The purpose of this study is to evaluate whether the administration of propranolol is safe and is able to reduce the incidence of blindness by suppressing the neovascular phase of ROP compared to a control group receiving conventional laser therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Infants who have been screened for ROP (≤ 32 weeks gestation) who develop Stage 2 ROP in zone II without plus.
2. Informed Consent from a parent

Exclusion Criteria:

1. Newborns with one or more of the following conditions at the enrollment in the study:

   * Heart failure.
   * Recurrent episodes of bradycardia (Heart rate less than 90 bpm).
   * Atrio-ventricular block (second or third degree).
   * Significant congenital heart anomaly, not including patent ductus arteriosus, patent foramen ovale or small ventricular septal defect.
   * Hypotension.
   * Renal failure.
   * Cerebral hemorrhage.
   * Other diseases which contraindicate the use of beta-blockers
2. Newborns with ROP stages more advances than Stage 2 in zone II without plus.
3. Informed Consent from a parent refused. This will mean that an infant automatically will receive standard laser therapy. No data will be used from an infant without Informed Consent.

Ages: 22 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2010-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The primary aim is to evaluate the safety of propranolol administration | Three months

SECONDARY OUTCOMES:
The secondary aim is to evaluate the efficacy of treatment with propranolol for reducing blindness and retinal detachment in newborns with ROP | six months from the beginning of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Luca Filippi, M.D., Principal Investigator — Azienda Ospedaliero-Universitaria A. Meyer, Firenze, Italy
Locations (2):
- Italy (2):
  - Neonatal Intensive Care Unit - Azienda Ospedaliero-Universitaria Meyer, Florence
  - Neonatal Intensive Care Unit - Fondazione IRCCS Cà Granda, Ospedale Maggiore Policlinico, Milan

REFERENCES:
- [Background] Filippi L, Cavallaro G, Fiorini P, Daniotti M, Benedetti V, Cristofori G, Araimo G, Ramenghi L, La Torre A, Fortunato P, Pollazzi L, la Marca G, Malvagia S, Bagnoli P, Ristori C, Dal Monte M, Bilia AR, Isacchi B, Furlanetto S, Tinelli F, Cioni G, Donzelli G, Osnaghi S, Mosca F. Study protocol: safety and efficacy of propranolol in newborns with Retinopathy of Prematurity (PROP-ROP): ISRCTN18523491. BMC Pediatr. 2010 Nov 18;10:83. doi: 10.1186/1471-2431-10-83. PMID 21087499
- [Derived] Filippi L, Cavallaro G, Bagnoli P, Dal Monte M, Fiorini P, Donzelli G, Tinelli F, Araimo G, Cristofori G, la Marca G, Della Bona ML, La Torre A, Fortunato P, Furlanetto S, Osnaghi S, Mosca F. Oral propranolol for retinopathy of prematurity: risks, safety concerns, and perspectives. J Pediatr. 2013 Dec;163(6):1570-1577.e6. doi: 10.1016/j.jpeds.2013.07.049. Epub 2013 Sep 18. PMID 24054431
- See also: Drug information — http://druginfo.nlm.nih.gov/